CLINICAL TRIAL: NCT06196125
Title: Ventilation dIstribution and effeCt of posTural Lateralization On Traumatic Lung injuRY: a Physiological Study
Acronym: VICTORY
Status: Active, not recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 23-231
Record Dates: First submitted 2023-12-23; First posted 2024-01-09 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Trauma Chest; Mechanical Ventilation
Keywords: chest trauma; mechanical ventilation; positional changes
MeSH Terms: conditions — Thoracic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intubated mechanically ventilated patients with thoracic trauma.: Intubated and mechanically ventilated patients with thoracic trauma (with at least 2 rib fractures with or without chest tube), who are in spontaneous/ partially assisted breathing phase.
  Interventions: Other: Four body positions

INTERVENTIONS:
Other: Four body positions — Physiological characteristics such as ventilation distribution and lung aeration patterns recorded by the electrical impedance tomography signals and ultrasound imaging will be measured when patients are in a initial supine position, then turned into a lateral positioning on each side then back in supine positioning.

SUMMARY:
This is a single-center, prospective, physiological study.

The study will enroll the traumatic lung injury patient who has at least 2 rib fractures requiring mechanical ventilation being on partially assisted breathing mode and on activity as tolerated (AAT) order with or without C-collar. Once being confirmed to meet the inclusion criteria, the research team will apply the EIT on the patient and start recording as well as perform lung ultrasound in the specific areas of interest in the selected time points of the study. The MV ventilator setting and some vital sign data will be also collected at selected time points of study. The EIT will continuously record from 5 minutes when patient is on supine position, then the investigators will turn patient using positioning wedge pillow to the sides with 30-minute EIT recording each side, lastly, the investigators will turn patient back to supine and continuously record for 30 minutes. The study will use the same protocol to perform in 3 different settings of mechanical ventilation (weaning process) i.) during partially assisted breathing, ii.) during high setting of spontaneous breathing and iii.) during low setting of spontaneous breathing.

DETAILED DESCRIPTION:
This study will be conducted while the patient is partially assisted on a breathing machine and have been clinically indicated to mobilize as tolerated while in the weaning process in the ICU.

The investigators will use EIT to visualize where air goes in the patient's lungs and lung ultrasonography to visualize lung inflation in specific areas. EIT is a measurement often used in the ICU since it allows easy visualization and is a non-invasive technique. The sensors measure electrical current changes during inspiration and expiration and will not cause any pain or radiation concerns. The EIT belt (3-cm diameter) will be placed around the chest without causing adverse event/discomfort/pain to the injured thorax area and recording will occur for 5 minutes during the first supine position, then 30 minutes for each side of left and right lateral position using the 30 Degree wedge pillow to support. The pillow is routinely applied to every ICU patient when eligible to be positioned on their side. As routine practice, patients are turned on each side every 2 hours to prevent pressure sores. Lastly, the investigators will do a final 30-minute recording when the patient is turned back onto their back. The duration of study will be approximately 95 minutes per session, which includes placing the patient in the four positions (on the back, the left side, the right side and returning to the back). The investigators will perform the same protocol at three different times when they are at different stages of weaning off the breathing machine: i) during partially assisted breathing, ii.) during a high setting of spontaneous breathing and iii.) during low setting of spontaneous breathing). These 3 breathing machine's settings indicate the patient is on the pathway of weaning off the breathing machine. The total study hours will be 4.75 hours (3 sessions) and each breathing machine's setting will be adjusted by clinical team over time. The investigators will proceed with the measurements only with agreement from the clinical team. The investigators will analyze the data collected offline with a dedicated software afterwards.

This study may require arterial blood gas analysis at baseline and after the procedure, only if there is an arterial line in place. The information from the sample provides the investigator the status of participant's breathing and breathing machine settings. It allows for any appropriate adjustments to the breathing machine. After these study procedures are completed, data will also be collected from the participant's chart and combined with relevant information from the breathing machine settings and vital functions at each stage of position changes. Confidentiality will be maintained throughout the entire study.

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥ 18 years
2. Traumatic lung injury with at least 2 rib fractures with or without chest tube and requiring mechanical ventilation
3. On any mode of ventilation including partially assisted breathing mode
4. With an "activity as tolerated (AAT) order" with or without C-collar

Exclusion Criteria:

1. Refusal of consent
2. Palliative or end of life condition
3. Contraindication to EIT placement: pacemaker/defibrillator implantation, burns at the area of EIT placement
4. Vasopressor: greater than 0.4 mcg/kg/min of norepinephrine infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be selected from intensive care units.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Difference in ventilation distribution (%) | 4.75 hours
  The primary endpoint is to study the difference of ventilation distribution (%) during different stages of spontaneous breathing/partially assisted breathing among four different body positions (supine 1, lateral 1, lateral 2, supine 2).
Difference in end expiratory lung volume (mL) | 4.75 hours
  The primary endpoint is to study end expiratory lung volume (EELV) in mL during different stages of spontaneous breathing/partially assisted breathing among four different body positions (supine 1, lateral 1, lateral 2, supine 2).

SECONDARY OUTCOMES:
Patterns of ventilation distribution. | 95 minutes
  To study the patterns of ventilation distribution and end expiratory lung volume during different stages of spontaneous breathing/partially assisted breathing on each position over period of time.
Correlation between ventilation distribution and lung aeration patterns. | 95 minutes
  Physiological characteristics: ventilation distribution recorded by electrical impedance tomography and ultrasound guidance during body position changes, correlation with body position changes over period of time, correlation with details of traumatic lung injury and correlation with mechanical ventilation days and Intensive care unit length of stay.
Quantify Pendelluft in different body positions | 95 minutes
  We would like to use electrical impedance tomography - a non-invasive and informative tool to study the ventilation distribution and the Pendelluft during spontaneous breathing or assisted ventilation during body position changes in traumatic lung injury patient.
Correlation of various traumatic lung injuries to ventilation distribution. | 95 minutes
  To identify the correlation among details of traumatic lung injury (type, location, number of rib fracture, side of rib fracture) with ventilation distribution, lung aeration patterns and effect of positional changes through ultrasound and electrical impedance tomography data.
Correlation of duration of mechanical ventilation to lung aeration patterns. | 95 minutes
  To identify the correlation of the previous duration of mechanical ventilation (from date of initiating mechanical ventilation to enrolment), with the result of ventilation distribution and lung aeration patterns from the effect of positional changes.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, MD, Principal Investigator — St. Michael's hospital, Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Electrical impedance tomography images and ultrasound images may be shared with no participant identification.